CLINICAL TRIAL: NCT06447168
Title: Prospective Non-interventional, Phase IV Multicentre Study to Assess the Effectiveness, Safety and Tolerability of Elafibranor 80 mg/Day in Participants With Primary Biliary Cholangitis Receiving Treatment in a Real-world Setting.
Brief Title: A Study Observing Everyday Effectiveness and Safety of the Drug Elafibranor in Participants With Primary Biliary Cholangitis Who Are Receiving Ongoing Treatment
Acronym: ELFINITY
Status: Recruiting | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: CLIN-60190-461
Record Dates: First submitted 2024-06-03; First posted 2024-06-06 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Primary Biliary Cholangitis
MeSH Terms: conditions — Liver Cirrhosis, Biliary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will collect information from participants with Primary Biliary Cholangitis (PBC) as they use the drug elafibranor in real world setting.

PBC is a progressive rare liver disease in which tubes in the liver called bile ducts are damaged.

The liver damage in PBC may lead to scarring (cirrhosis). PBC may also be associated with multiple symptoms including pruritus (itching) and fatigue. Many patients with PBC may require liver transplant or may die if the disease progresses and a liver transplant is not done.

In this study the main aim is to observe the effectiveness, safety and tolerability of elafibranor in participants with PBC who are receiving treatment in real world setting. The total study duration for each participants will be 60 months (approximately 5 years).

ELIGIBILITY:
Inclusion Criteria:

* Participant has provided written informed consent and agrees to comply with the study protocol.
* Participant with PBC diagnosis.
* Participant for whom the treating physician has decided to start or participants who are currently receiving treatment with commercialized elafibranor.
* If a participant has a caregiver who agrees to complete the caregiver questionnaires, an informed consent should be collected from the caregiver before any data is collected.

Exclusion Criteria:

* Participant is currently participating or, plans to participate in an investigational drug study or medical device study containing active substance.
* Participant with known hypersensitivity to the product or to any of its excipients.
* Participant with mental instability or incompetence, such that the validity of informed consent or ability to be compliant with the study is uncertain.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with PBC for whom the treating physician has decided to start treatment with elafibranor 80 mg/day, as recommended in the approved indication.
Sampling Method: Non-Probability Sample
Enrollment: 424 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2032-07-15 (Estimated); Study Completion 2032-07-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with response to treatment | At month 6
  Defined as alkaline phosphatase (ALP) <1.67 x upper limit of normal (ULN) and total bilirubin (TB) ≤ULN and ALP decrease ≥15% from baseline.

SECONDARY OUTCOMES:
Percentage of participants with normalization of ALP levels | Up to 60 months following enrollment, based on routine physician follow-up visit
Percentage of participants with response to treatment | Up to 60 months following enrollment, based on routine physician follow-up visits
  Defined as ALP<1.67 x ULN and TB≤ULN and ALP decrease ≥15% from baseline.
Change from baseline in liver function parameters: Serum levels of alanine aminotransferase (ALT) | Up to 60 months following enrollment, based on routine physician follow-up visit
Change from baseline in liver function parameters: Serum levels of Aspartate aminotransferase (AST) | Up to 60 months following enrollment, based on routine physician follow-up visit
Change from baseline in liver function parameters: Serum levels of Gamma-glutamyl transferase (GGT) | Up to 60 months following enrollment, based on routine physician follow-up visit
Change from baseline in liver function parameters: Serum levels of TB | Up to 60 months following enrollment, based on routine physician follow-up visit
Change from baseline in liver function parameters: Conjugated (direct) bilirubin | Up to 60 months following enrollment, based on routine physician follow-up visit
Change from baseline in liver function parameters: Serum levels of creatinine | Up to 60 months following enrollment, based on routine physician follow-up visit
Change from baseline in liver function parameters: Serum levels of albumin | Up to 60 months following enrollment, based on routine physician follow-up visit
Change from baseline in pruritus based on PBC Itch score | Up to 60 months following enrollment, based on routine physician follow-up visit
  The PBC Itch score is a simple, self-administered Patient Reported Outcome (PRO) questionnaire that measures itch intensity. It uses 7-day recall periods and asks participants to rate the intensity of their worst itch over the past 7-day period on an 11-point scale ranging from 0 (no itch) to 10 (worst itch imaginable).
Change from baseline in fatigue based on functional assessment of chronic illness therapy-fatigue (FACIT-Fatigue) scale | Up to 60 months following enrollment, based on routine physician follow-up visit
  The FACIT-Fatigue is a 13-item measure that assesses self-reported fatigue and its impact upon daily activities and function. It is a subset of the longer (47-item) Functional Assessment of Cancer Therapy - Anemia (FACT-An), which includes the 27-item FACT-G and a 20-item subscale addressing additional concerns associated with the anemia of cancer and its treatment. This 20-item subscale, referred to as the anemia subscale, is comprised of 13-items that assess fatigue and its impact (the FACIT-Fatigue) and, 7 additional symptoms associated with anemia (e.g. shortness of breath, headache). participants rate their symptoms over the preceding seven days on a verbal response scale, the options range from 'not at all' / 'a little bit' / 'somewhat quite a bit' / very much'.
Change from baseline in sleep based on Pittsburgh sleep quality index (PSQI) | Up to 60 months following enrollment, based on routine physician follow-up visit
  The PSQI was designed to evaluate overall sleep quality in the psychiatric disorders associated with sleep disturbances. Each of the questionnaire's 19-self-reported items belongs to one of seven subcategories: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. Five additional questions rated by the respondent's roommate or bed partner are included for clinical purposes and are not scored.
Change from baseline in Quality Of Life (QoL) based on PBC-40 questionnaire | Up to 60 months following enrollment, based on routine physician follow-up visit
  The PBC-40 is a validated, PBC-specific, health-related Quality Of Life (QoL) questionnaire with 40 questions that assesses symptoms across six domains: fatigue, emotional and social, cognitive function, general symptoms and itch. Participants respond on a verbal response scale, depending on the section options range from 'never' / 'not at all' / 'strongly disagree' to 'always' / 'very much'/ 'strongly agree'. Five items (3/3 in the itch domain and 2/10 in the social domain) also include a 'does not apply' option. A score for each domain is provided (but a total score is not calculated), with each verbal response scale correlating to a score of 1-5 per item (0-5 on items with a 'does not apply' option) with 5 being the most affected.
Change from baseline in QoL based on 5-Dimensional Itch scale (5-D Itch, also known as 5-D pruritus scale) | Up to 60 months following enrollment, based on routine physician follow-up visit
  The 5-D Itch scale assesses symptoms in terms of five domains: degree, duration, direction, disability and distribution. It is a 1 to 5 scale, with 5 being the most affected.
Change from baseline in liver stiffness | Up to 60 months following enrollment, based on routine physician follow-up visit
  Measured by transient elastography (FibroScan®) and enhanced liver fibrosis (ELF) test
Event free survival | From baseline to up to 60 months
  Event free survival from first intake of commercialized elafibranor treatment as prescribed by physician to the first occurrence of any of the following clinical outcome events: (1) death, (2) liver transplant, and (3) liver decompensation.
Percentage of participants experiencing Adverse Events (AEs), Adverse Events of Special Interests (AESIs) and special situations (SS). | From baseline to up to 60 months
  An Adverse event (AE) is any untoward medical occurrence, temporally associated with the use of study intervention, whether or not related to the study intervention. AESIs are AEs that may not be serious but are of special importance to a particular drug or class of drugs.
Participant's satisfaction on treatment | Up to 60 months following enrollment, based on routine physician follow-up visit
  Measured by treatment satisfaction questionnaire for medication (TSQM). The TSQM (version 1.4) has 14 questions divided into 4 subscales: effectiveness (items 1 to 3), side effects (items 4 to 8), convenience (items 9 to 11), and global satisfaction (items 12 to 14).
Participant's adherence to treatment | Up to 60 months following enrollment, based on routine physician follow-up visit
  Adherence to the treatment will be measured based on the participant report of missed doses every month.
Percentage of participants with clinically significant changes in laboratory parameters | Up to 60 months following enrollment, based on routine physician follow-up visit
  Percentage of participants with clinically significant change in laboratory parameters (blood chemistry, hematology and coagulation) will be reported. The clinical significance will be graded by the investigator.
Percentage of participants with clinically significant changes in physical examination | Up to 60 months following enrollment, based on routine physician follow-up visit
  Clinically significant changes in physical examination will be reported. The clinical significance will be graded by the investigator.
Percentage of participants developing clinically significant changes in vital signs | Up to 60 months following enrollment, based on routine physician follow-up visit
  Clinically significant changes in vital signs will be reported. The clinical significance will be graded by the investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (58):
- United States (19):
  - Southern California Research Center, Coronado, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California Davis Medical Center, Sacramento, California
  - South Denver Gastroenterology,P.C., Englewood, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Schiff Center for Liver Diseases - University of Miami, Miami, Florida
  - Beth Israel Deaconess Medical Center, Liver Research Center, Boston, Massachusetts
  - Virtua Center for Liver Disease - Cherry Hill, Cherry Hill, New Jersey
  - Northwell Health Inc, Center for Liver Disease and Transplantation, Manhasset, New York
  - UNC Hospitals, The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Liver Center of Texas, Dallas, Texas
  - Baylor College of Medicine - Advanced Liver Therapies, Houston, Texas
  - Gastro health & Nutrition, Katy, Texas
  - Intermountain Medical Center, Murray, Utah
  - Bon Secours Richmond Community Hospital LLC. d/b/a Bon Secours Liver Institute of Richmond, Richmond, Virginia
  - Virginia Commonwealth University Medical Center - West Hospital, Richmond, Virginia
  - Velocity Clinical Research, Seattle, Washington
- Austria (2):
  - Medizinische Universitaetsklinik Graz, Graz
  - Medical University Innsbruck, Innsbruck
- Canada (4):
  - University of Calgary, Calgary
  - London Health Sciences Centre (LHSC) - University Hospital, London
  - The Ottawa Hospital - General Campus, Ottawa
  - (G.I.R.I) GI Research Institute Foundation, Vancouver
- Germany (8):
  - Charite Universitatsmedizin Berlin, Berlin
  - DRK Kliniken Berlin Mitte, Berlin
  - Klinikum der Johann Wolfgang Goethe-Universitaet, Frankfurt
  - Studiengesellschaft BSF, Halle
  - Gastroenterologsiche Studiengesellschaft Herne, Herne
  - Universitaet des Saarlandes, Homburg
  - Universitaetsklinikum Leipzig, Leipzig
  - Hospital of the Merciful Brothers Trier, Trier
- Greece (5):
  - General Hospital of Athens Laiko, Athens
  - University Hospital of Heraklion, Heraklion
  - University General Hospital of Larissa, Larissa
  - University General Hospital of Patras, Pátrai
  - Ippokratio General Hospital of Thessaloniki, Thessaloniki
- Italy (7):
  - ASST-Ospedale Papa Giovanni XXIII, Bergamo
  - Ospedale Garibaldi Nesima, Catania
  - Universita Degli Studi Di Firenze - Azienda Ospedaliero-Universitaria Careggi (AOUC), Florence
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Ospedale Maggiore Della Carita, Novara
  - A. Gemelli University Hospital, Catholic University of the Sacred Heart, Roma
  - Fondazione Policlinico Universitario Campus Bio-Medico, Roma
- United Arab Emirates (4):
  - Clemenceau Medical Center Hospital, Dubai
  - Mediclinic Airport Road Hospital, Dubai
  - Rashid Hospital, Dubai
  - Sheikh Shakhbout Medical City, Dubai
- United Kingdom (9):
  - Aberdeen Royal Infirmary NHS Grampian Grampian Health Board, Aberdeen
  - Belfast Health and Social Care Trust - Royal Victoria Hospital, Belfast
  - Queen Elizabeth Hospital Birmingham - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Bradford Royal Infirmary - Bradford Teaching Hospitals NHS Foundation, Bradford
  - Hull Royal Infirmary - Hull University Teaching Hospitals NHS Trust, Hull
  - King's College Hospital NHS Foundation Trust, London
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust - Freeman Hospital, Newcastle
  - Queen's Medical Centre - Nottingham University Hospitals NHS Trust, Nottingham
  - John Radcliffe Hospital - Oxford University Hospitals NHS Foundation Trust, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications.
  Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and/or EU.
Access Criteria: Further details on Ipsen's sharing criteria and process for sharing are available here (https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/).
URL: https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/